CLINICAL TRIAL: NCT00379821
Title: A Longitudinal Study of Chloroquine as Monotherapy or in Combination With Artesunate, Azithromycin or Atovaquone-Proguanil to Treat Malaria in Children in Blantyre, Malawi
Brief Title: Chloroquine Alone or in Combination for Malaria in Children in Malawi
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0022
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Results first posted 2011-07-27 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Plasmodium Falciparum Infection
Keywords: chloroquine, malaria, Plasmodium falciparum, Malawi, children
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — atovaquone, proguanil drug combination; Artesunate; Azithromycin; Chloroquine

ARMS (4):
- CQ Monotherapy (Experimental): N=160: treat with Chloroquine (CQ) alone.
  Interventions: Drug: Chloroquine
- CQ plus atovaquone proguanil (Experimental): N=160: treat with CQ plus atovaquone proguanil.
  Interventions: Drug: Atovaquone-proguanil; Drug: Chloroquine
- CQ plus artesunate (Experimental): N=160: treat with CQ plus artesunate.
  Interventions: Drug: Artesunate; Drug: Chloroquine
- CQ plus azithromycin (Experimental): N=160: treat with CQ plus azithromycin.
  Interventions: Drug: Azithromycin; Drug: Chloroquine

INTERVENTIONS:
Drug: Atovaquone-proguanil — Atovaquone-proguanil: once a day for 3 days, Pediatric tablet: 62.5 mg/25 mg, Full strength tablet: 250 mg/100 mg
  Arms: CQ plus atovaquone proguanil
Drug: Artesunate — Artesunate: 4mg/kg once a day for 3 days, 50 mg tablet
  Arms: CQ plus artesunate
Drug: Azithromycin — Azithromycin 30 mg/kg once a day for 3 days, 200 mg/5cc suspension
  Arms: CQ plus azithromycin
Drug: Chloroquine — Chloroquine: 10 mg/kg on days 0 and 1, 5 mg/kg/day on day 2, 100 mg tablet.

SUMMARY:
Malaria is a sickness caused by a germ that can get into a person's body when a mosquito bites them. It can cause fever, headache, body aches and weakness. It can even cause death, especially in children. When malaria is treated with the appropriate medicine(s), it can be cured completely. The purpose of this study is to find out if it is better to use chloroquine alone or in combination with another drug to most effectively treat malaria. About 640 children with malaria, aged 6 months to 5 years of age, from the Blantyre Malaria Project Research Clinic at the Ndirande Health Center in Malawi will be in the study. They will be treated with either chloroquine alone or a combination of chloroquine plus another medication (azithromycin or artesunate or atovaquone-proguanil) every time they get malaria for a year. Blood samples will be collected and tested at least every 4 weeks. Participants will be involved in the study for 1 year.

DETAILED DESCRIPTION:
Combination therapy is becoming the mainstay of malaria treatment. In general, the goal of combination therapy is to treat resistant infections successfully and to prevent the emergence and spread of resistance. The antimalarial combination therapies currently in use were not designed based on optimal pairing of drugs to deter the development and spread of parasite resistance to the individual partner drugs in settings of high malaria transmission. Careful studies are needed to identify the pharmacokinetic and pharmacodynamic properties of drug combinations that will deter resistance and prolong the useful therapeutic life of the next generation of antimalarial drug combinations. Current in vivo methods for measuring antimalarial drug efficacy in high-transmission areas use a 14 or 28-day follow-up period, but a single episode study misses several critical factors in assessing the efficacy and impact of antimalarial treatment. When follow-up is extended beyond 28 days, more cases of apparent resistance or treatment failure are found. Single-episode studies cannot assess the impact of therapy on the incidence of malaria over time. These limitations of standard in vivo studies have led the investigators to advocate longitudinal studies of drug efficacy. In addition to measuring efficacy of individual treatments, longitudinal studies measure sustained efficacy with repeated use of the same regimen over time, a scenario that more accurately reflects the real-life use of anti-malarial medication. The primary outcome of interest is the incidence of malaria episodes, as well as the secondary outcomes of anemia and severe malaria, are all highly relevant to public health policy-makers, as they reflect not only the burden of disease but also the utilization of health resources. Longitudinal studies also permit assessment of how pharmacokinetic properties of drugs affect the incidence of treatment episodes. This is a randomized, open-label, longitudinal drug efficacy trial. Participants will include 640 children, aged 6 months to 5 years, who are found to have uncomplicated malaria at the Blantyre Malaria Project Research Clinic at the Ndirande Health Centre in Blantyre, Malawi. After enrollment, participants will be randomized to one of four treatment arms: chloroquine alone or chloroquine in combination with artesunate, atovaquone-proguanil (AP), or azithromycin. The treatment outcome will be assessed through a standard 28-day efficacy study. Participants will subsequently be evaluated every 4 weeks and encouraged to return to the study clinic any time they are ill during the course of one year. If a new episode of uncomplicated malaria is diagnosed, the participant will receive the same therapy as assigned on enrollment. Polymerase chain reaction-corrected 28-day efficacy will be evaluated for each treatment episode. The primary study objective is to compare annual incidence of malaria clinical episodes. Secondary objectives are to: assess anti-malarial drug efficacy at first administration, by treatment arm; assess anti-malarial drug efficacy during subsequent episodes of malaria, by treatment arm; measure prevalence of chloroquine resistant parasites during the trial, by treatment arm; assess effect of each treatment arm on anemia at the end of study participation; assess safety of these drugs with repeated use; determine the chloroquine blood levels at which chloroquine sensitive and resistant parasites are able to cause infection; assess the effect of population movements on the risk of malaria infection; and assess the spatial patterns and the environmental determinants of malaria infection. Participants will be involved in study rela

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged greater than or equal to 6 months to 5 years presenting to Ndirande Health Centre with signs or symptoms consistent with malaria including, but not limited to, one or more of the following:

  1. fever at the time of evaluation (axillary temperature greater than or equal to 37.5 degrees Celsius by digital thermometer)
  2. report of fever within the last two days
  3. clinically profound anemia (conjunctival or palmar pallor)
  4. headache
  5. body aches
  6. abdominal pain
  7. decreased intake of food or fluids
  8. weakness
* Weight greater than or equal to 5kg.
* Positive malaria smear for P. falciparum mono-infection with parasite density 2,000-200,000/mm^3.
* Planning to remain in the study area for 1 year.
* Willingness to return for four-weekly routine visits, as well as unscheduled sick visits.
* Parental/guardian consent for each participant.

Exclusion Criteria:

* Signs of severe malaria: One or more of the following:

  1. hemoglobin less than or equal to 5 g/dL
  2. prostration
  3. respiratory distress
  4. bleeding
  5. recent seizures, coma or obtundation (Blantyre coma score < 5)
  6. inability to drink
  7. persistent vomiting
* Known allergy or history of adverse reaction to chloroquine (CQ), artesunate, azithromycin, erythromycin or atovaquone-proguanil (AP)
* Chronic medication with any antibiotic or anti malarial medication
* Previous enrollment in this study
* Alanine aminotransferase (ALT) more than 5x the upper limit of normal or creatinine greater than 3x the upper limit of normal
* Evidence of chronic disease or physical stigmata of severe malnutrition (i.e., loss of muscle mass or subcutaneous tissue, edema, or skin or hair findings consistent with severe malnutrition)

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 640 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Blantyre Malaria Project - Ndirande Health Centre, Blantyre, Blantyre, Malawi

REFERENCES:
- [Background] Laufer MK, Thesing PC, Dzinjalamala FK, Nyirenda OM, Masonga R, Laurens MB, Stokes-Riner A, Taylor TE, Plowe CV. A longitudinal trial comparing chloroquine as monotherapy or in combination with artesunate, azithromycin or atovaquone-proguanil to treat malaria. PLoS One. 2012;7(8):e42284. doi: 10.1371/journal.pone.0042284. Epub 2012 Aug 17. PMID 22912697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children who were brought to the Ndirande Health Centre with symptoms suggestive of malaria were recruited from February 19, 2007 to August 13, 2008.
Groups:
- Chloroquine Plus Artesunate: Participants receive chloroquine (CQ) at 10 mg/kg on days 0 and 1, and 5 mg/kg/day on day 2; plus Artesunate at a dose of 4 mg/kg once a day for 3 days.
- Chloroquine Plus Atovaquone-Proguanil: Participants receive CQ at 10 mg/kg on days 0 and 1, and 5 mg/kg/day on day 2; plus Atovaquone-Proguanil (AP) once a day for 3 days dosed as follows: 5-8 kg, 2 pediatric tablet (PT, 62.5 mg/25mg); 9-10 kg, 3 PT; 11-20 kg, 1 full strength tablet (FST, 250mg/100 mg); 21-30 kg 2 FST; >30 kg, 3 FST.
- CQ Plus Azithromycin: Participants receive CQ at 10 mg/kg on days 0 and 1, and 5 mg/kg/day on day 2; plus Azithromycin 30 mg/kg once a day for 3 days.
- CQ Monotherapy: Participants receive CQ at 10 mg/kg on days 0 and 1, and 5 mg/kg/day on day 2.
Period: Overall Study
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Started | 160 | 160 | 160 | 160
Completed | 87 | 71 | 93 | 81
Not Completed | 73 | 89 | 67 | 79

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy | Total
Number analyzed (Participants) | 160 | 160 | 160 | 160 | 640
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 160 | 160 | 160 | 160 | 640
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.7 (1.2) | 2.7 (1.2) | 2.8 (1.1) | 2.7 (1.2) | 2.7 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 82 | 73 | 77 | 302
  Male | 90 | 78 | 87 | 83 | 338
Region of Enrollment [Number; unit: participants]
  Malawi | 160 | 160 | 160 | 160 | 640

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinical Malaria Episodes Per Year of Follow-up
Description: Clinical malaria episode was defined as at least one symptom of malaria and a positive malaria smear. The number of clinical malaria episodes (not including the initial malaria episode) reported by participants during follow up is presented as the number per Person Years at Risk (PYAR).
Time Frame: 1 year
Population: The intention to treat (ITT) population was used for the primary outcome.
Measure: Number; unit: Episodes per PYAR
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 157 | 155 | 160 | 156
Episodes per PYAR | 0.61 | 0.68 | 0.64 | 0.59
Statistical Analysis 1: Comparison: Chloroquine Plus Artesunate vs CQ Monotherapy; Number of clinical malaria episodes per PYAR was compared using Poisson regression assuming null hypothesis that the number of malaria episodes are the same in both groups; Test type: Superiority or Other; p = 0.8097, Poisson regression — The a priori threshold for statistical significance is 0.05/3; No adjustments; Risk Ratio (RR) = 1.0413, 95% CI 2-sided [0.7497 to 1.4463], Standard Error of Mean 0.1746 — The denominator for the risk ratio is the CQ Monotherapy arm
Statistical Analysis 2: Comparison: Chloroquine Plus Atovaquone-Proguanil vs CQ Monotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3767, Poisson regression — The a priori threshold for statistical significance is 0.05/3; No adjustments; Risk Ratio (RR) = 1.1623, 95% CI 2-sided [0.8333 to 1.6211], Standard Error of Mean 0.1973 — The denominator for the risk ratio is the CQ Monotherapy arm
Statistical Analysis 3: Comparison: CQ Plus Azithromycin vs CQ Monotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6277, Poisson regression — The a priori threshold for statistical significance is 0.05/3; No adjustments; Risk Ratio (RR) = 1.0707, 95% CI 2-sided [0.7708 to 1.4872], Standard Error of Mean 0.1795 — The denominator for the risk ratio is the CQ Monotherapy arm

2. Secondary Outcome: Number of Participants With Day 28 Adequate Clinical and Parasitologic Response in Each Treatment Arm
Description: Adequate clinical and parasitologic response (ACPR) was defined as the absence of parasitemia at Day 28 and without previously meeting any of the criteria of early treatment or late clinical failure.
Time Frame: Day 28 of initial malaria episode (Episode 0)
Population: This analysis was per protocol, which excludes participants who did not have p. falciparum or who did not receive all 3 doses of treatment.
Measure: Number; unit: Participants
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 144 | 133 | 138 | 135
Participants | 143 | 133 | 137 | 135

3. Secondary Outcome: Number of Participants With Day 28 Adequate Clinical and Parasitologic Response in Each Treatment Arm
Description: as for outcome 2
Time Frame: Day 28 of first subsequent malaria episode (Episode 1)
Population: This analysis was per protocol, which includes participants who had at least 1 subsequent malaria episode, but excludes participants who did if that episode was not caused by p. falciparum or if the participant did not receive all 3 doses of treatment for the first subsequent episode.
Measure: Number; unit: Participants
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 46 | 42 | 39 | 41
Participants | 46 | 42 | 37 | 39

4. Secondary Outcome: Number of Participants With Day 28 Adequate Clinical and Parasitologic Response in Each Treatment Arm
Description: as for outcome 2
Time Frame: Day 28 of second subsequent malaria episode (Episode 2)
Population: This analysis was per protocol, which which includes participants who had at least 2 subsequent malaria episodes, but excludes participants if the second episode was not caused by p. falciparum or if the participant did not receive all 3 doses of treatment for the second episode.
Measure: Number; unit: Participants
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 17 | 14 | 12 | 6
Participants | 17 | 14 | 12 | 6

5. Secondary Outcome: Number of Participants With Day 28 Adequate Clinical and Parasitologic Response in Each Treatment Arm
Description: as for outcome 2
Time Frame: Day 28 of third subsequent malaria episode (Episode 3)
Population: This analysis was per protocol, which includes participants who had at least 3 subsequent malaria episodes, but excludes participants if the third episode was not caused by p. falciparum or if the participant did not receive all 3 doses of treatment for the third episode.
Measure: Number; unit: Participants
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 4 | 4 | 7 | 1
Participants | 4 | 4 | 6 | 0

6. Secondary Outcome: Number of Participants With Day 28 Adequate Clinical and Parasitologic Response in Each Treatment Arm
Description: as for outcome 2
Time Frame: Day 28 of fourth subsequent malaria episode (Episode 4)
Population: This analysis was per protocol, which includes participants who had 4 subsequent malaria episodes, but excludes participants if the fourth episode was not caused by p. falciparum or if the participant did not receive all 3 doses of treatment for the fourth episode.
Measure: Number; unit: Participants
Groups:
- Chloroquine Plus Atovaquone-Proguanil: Subjects receive CQ at 10 mg/kg on days 0 and 1, and 5 mg/kg/day on day 2; plus Atovaquone-Proguanil (AP) once a day for 3 days dosed as follows: 5-8 kg, 2 pediatric tablet (PT, 62.5 mg/25mg); 9-10 kg, 3 PT; 11-20 kg, 1 full strength tablet (FST, 250mg/100 mg); 21-30 kg 2 FST; >30 kg, 3 FST.
- CQ Plus Azithromycin: Subjects receive CQ at 10 mg/kg on days 0 and 1, and 5 mg/kg/day on day 2; plus Azithromycin 30 mg/kg once a day for 3 days.
Arm/Group | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

7. Secondary Outcome: Number of Cases of Severe Malaria in Each Treatment Arm
Description: A case of severe malaria included one or more of the following: Hemoglobin ≤5 g/dL; prostration; respiratory distress; bleeding; recent seizures, coma or obtundation (Blantyre coma score < 5); inability to drink, or persistent vomiting. All cases were then adjudicated by a panel of investigators prior to analysis.
Time Frame: 1 Year
Population: The safety cohort includes all participants.
Measure: Number; unit: Cases of severe malaria
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 160 | 160 | 160 | 160
Cases of severe malaria | 0 | 2 | 2 | 6

8. Secondary Outcome: Mean Hemoglobin at the Last Study Visit in Each Treatment Arm for the Age Group of Participants 3 Years of Age or Younger.
Description: Hemoglobin values were assessed from blood collected at the last study visit at one year after enrollment. Group means are stratified by participants 3 years of age and under, and over 3 to 5 years of age.
Time Frame: 1 year
Population: The safety population includes all participants. The number of participants is limited to those who attended the final 1-year visit.
Measure: Mean (95% Confidence Interval); unit: Grams/Deciliter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 44 | 35 | 50 | 48
Grams/Deciliter | 11.6 [11.3 to 12.0] | 11.7 [11.4 to 12.0] | 12.2 [11.8 to 12.6] | 11.8 [11.4 to 12.1]

9. Secondary Outcome: Mean Hemoglobin at the Last Study Visit in Each Treatment Arm for the Age Group of Participants Greater Than 3 Years to 5 Years of Age.
Description: as for outcome 8
Time Frame: 1 year
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Grams/Deciliter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 39 | 34 | 40 | 29
Grams/Deciliter | 12.5 [12.1 to 12.8] | 12.3 [12.0 to 12.7] | 12.1 [11.8 to 12.3] | 12.5 [12.0 to 13.0]

10. Secondary Outcome: Mean Creatinine in Each Treatment Arm (Renal Function)
Description: Creatine values were assessed from blood draws at Day 0 and Day 14 of each malaria episode. Samples that were below the limit of detection were reported as 44.2 micromoles/liter, equivalent to the lower limit of detection.
Time Frame: Day 0 of initial malaria episode (Episode 0)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: Micromole/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 160 | 160 | 158 | 160
Micromole/Liter | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.3] | 44.2 [44.2 to 44.2] | 44.3 [44.1 to 44.5]

11. Secondary Outcome: Mean Creatinine in Each Treatment Arm (Renal Function)
Description: as for outcome 10
Time Frame: Day 14 of initial malaria episode (Episode 0)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: Micromole/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 144 | 138 | 143 | 141
Micromole/Liter | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2]

12. Secondary Outcome: Mean Creatinine in Each Treatment Arm (Renal Function)
Description: as for outcome 10
Time Frame: Day 0 of first subsequent malaria episode (Episode 1)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: Micromole/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 54 | 49 | 47 | 52
Micromole/Liter | 43.9 [43.4 to 44.5] | 44.2 [44.2 to 44.3] | 43.7 [42.9 to 44.5] | 43.6 [42.7 to 44.4]

13. Secondary Outcome: Mean Creatinine in Each Treatment Arm (Renal Function)
Description: as for outcome 10
Time Frame: Day 14 of first subsequent malaria episode (Episode 1)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: Micromole/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 53 | 43 | 45 | 46
Micromole/Liter | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2]

14. Secondary Outcome: Mean Creatinine in Each Treatment Arm (Renal Function)
Description: as for outcome 10
Time Frame: Day 0 of second subsequent malaria episode (Episode 2)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: Micromole/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 17 | 15 | 18 | 9
Micromole/Liter | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2] | 46.4 [41.4 to 51.3]

15. Secondary Outcome: Mean Creatinine in Each Treatment Arm (Renal Function)
Description: as for outcome 10
Time Frame: Day 14 of second subsequent malaria episode (Episode 2)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: Micromole/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 17 | 14 | 16 | 8
Micromole/Liter | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2]

16. Secondary Outcome: Mean Creatinine in Each Treatment Arm (Renal Function)
Description: as for outcome 10
Time Frame: Day 0 of third subsequent malaria episode (Episode 3)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: Micromole/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 4 | 4 | 7 | 1
Micromole/Liter | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2] | 44.2

17. Secondary Outcome: Mean Creatinine in Each Treatment Arm (Renal Function)
Description: as for outcome 10
Time Frame: Day 14 of third subsequent malaria episode (Episode 3)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: Micromole/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 3 | 4 | 6 | 1
Micromole/Liter | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2] | 44.2 [44.2 to 44.2] | 44.2

18. Secondary Outcome: Mean Creatinine in Each Treatment Arm (Renal Function)
Description: as for outcome 10
Time Frame: Day 0 of fourth subsequent malaria episode (Episode 4)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: Micromole/Liter
Arm/Group | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin
Number analyzed (Participants) | 2 | 1
Micromole/Liter | 44.2 [44.2 to 44.2] | 44.2

19. Secondary Outcome: Mean Creatinine in Each Treatment Arm (Renal Function)
Description: as for outcome 10
Time Frame: Day 14 of fourth subsequent malaria episode (Episode 4)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: Micromole/Liter
Arm/Group | Chloroquine Plus Atovaquone-Proguanil
Number analyzed (Participants) | 1
Micromole/Liter | 44.2

20. Secondary Outcome: Mean Alanine Transaminase (ALT) in Each Treatment Arm (Hepatic Function)
Description: ALT values were assessed from blood draws at Day 0 and Day 14 of each malaria episode.
Time Frame: Day 0 of initial malaria episode (Episode 0)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: International Units/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 160 | 160 | 158 | 160
International Units/Liter | 27.2 [23.1 to 31.2] | 32.1 [25.7 to 38.4] | 27.5 [23.0 to 31.9] | 26.2 [23.1 to 29.3]

21. Secondary Outcome: Mean Alanine Transaminase (ALT) in Each Treatment Arm (Hepatic Function)
Description: ALT values were assessed from blood draws at Day 0 and Day 14 of each malaria episode.
Time Frame: Day 14 of initial malaria episode (Episode 0)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: International Units/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 144 | 138 | 143 | 142
International Units/Liter | 14.3 [13.5 to 15.2] | 16.2 [14.9 to 17.4] | 17.8 [15.5 to 20.1] | 15.5 [14.4 to 16.6]

22. Secondary Outcome: Mean Alanine Transaminase (ALT) in Each Treatment Arm (Hepatic Function)
Description: ALT values were assessed from blood draws at Day 0 and Day 14 of each malaria episode.
Time Frame: Day 0 of first subsequent malaria episode (Episode 1)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: International Units/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 54 | 49 | 47 | 52
International Units/Liter | 24.2 [19.9 to 28.6] | 21.7 [14.8 to 28.5] | 22.4 [17.9 to 27.0] | 25.3 [18.8 to 31.8]

23. Secondary Outcome: Mean Alanine Transaminase (ALT) in Each Treatment Arm (Hepatic Function)
Description: ALT values were assessed from blood draws at Day 0 and Day 14 of each malaria episode.
Time Frame: Day 14 of first subsequent malaria episode (Episode 1)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: International Units/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 53 | 43 | 45 | 46
International Units/Liter | 14.5 [13.2 to 15.9] | 14.2 [12.8 to 15.6] | 18.3 [14.1 to 22.5] | 17.2 [15.0 to 19.5]

24. Secondary Outcome: Mean Alanine Transaminase (ALT) in Each Treatment Arm (Hepatic Function)
Description: ALT values were assessed from blood draws at Day 0 and Day 14 of each malaria episode.
Time Frame: Day 0 of second subsequent malaria episode (Episode 2)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: International Units/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 17 | 15 | 18 | 9
International Units/Liter | 26.1 [17.9 to 34.2] | 23.0 [16.3 to 29.8] | 23.3 [12.3 to 34.2] | 23.5 [15.6 to 31.4]

25. Secondary Outcome: Mean Alanine Transaminase (ALT) in Each Treatment Arm (Hepatic Function)
Description: ALT values were assessed from blood draws at Day 0 and Day 14 of each malaria episode.
Time Frame: Day 14 of second subsequent malaria episode (Episode 2)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: International Units/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 17 | 14 | 16 | 8
International Units/Liter | 116 [0 to 333] | 14.7 [11.8 to 17.6] | 17.3 [9.8 to 24.8] | 16.3 [13.8 to 18.9]

26. Secondary Outcome: Mean Alanine Transaminase (ALT) in Each Treatment Arm (Hepatic Function)
Description: ALT values were assessed from blood draws at Day 0 and Day 14 of each malaria episode.
Time Frame: Day 0 of third subsequent malaria episode (Episode 3)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: International Units/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 4 | 4 | 7 | 1
International Units/Liter | 26.4 [18.0 to 34.8] | 20.7 [7.3 to 34.0] | 18.6 [12.6 to 24.5] | 16.2

27. Secondary Outcome: Mean Alanine Transaminase (ALT) in Each Treatment Arm (Hepatic Function)
Description: ALT values were assessed from blood draws at Day 0 and Day 14 of each malaria episode.
Time Frame: Day 14 of third subsequent malaria episode (Episode 3)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: International Units/Liter
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 3 | 4 | 6 | 1
International Units/Liter | 17.8 [0 to 44.3] | 13.6 [8.2 to 18.9] | 15.3 [8.7 to 21.8] | 14.3

28. Secondary Outcome: Mean Alanine Transaminase (ALT) in Each Treatment Arm (Hepatic Function)
Description: ALT values were assessed from blood draws at Day 0 and Day 14 of each malaria episode.
Time Frame: Day 0 of fourth subsequent malaria episode (Episode 4)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: International Units/Liter
Arm/Group | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin
Number analyzed (Participants) | 2 | 1
International Units/Liter | 27.3 [0 to 95.2] | 24.9

29. Secondary Outcome: Mean Alanine Transaminase (ALT) in Each Treatment Arm (Hepatic Function)
Description: ALT values were assessed from blood draws at Day 0 and Day 14 of each malaria episode.
Time Frame: Day 14 of fourth subsequent malaria episode (Episode 4)
Population: The safety population includes all participants who have laboratory results reported at the time point for the episode.
Measure: Mean (95% Confidence Interval); unit: International Units/Liter
Arm/Group | Chloroquine Plus Atovaquone-Proguanil
Number analyzed (Participants) | 1
International Units/Liter | 13.9

30. Secondary Outcome: Number of Participants in Each Treatment Arm Who Change From "Normal" to "Abnormal" on Any Questions of the Neurological Examination
Description: A basic age-appropriate neurological examination was conducted on Day 28 of each malaria illness episode and also at Days 112 and 224, and at 1 year. Subjects were were counted as a "change from 'normal' to 'abnormal' " if they had the 'normal' (or not-applicable) response for the initial day 28 exam and an 'abnormal' response at their last exam. If a subject did not have an exam at 1 year then the last available exam that was not associated with an illness episode (either Day 112 or 224) was used.
Time Frame: 1 Year
Population: Subjects who did not have an initial exam, or who did not have a subsequent exam at a routine visit are excluded.
Measure: Number; unit: Participants
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 132 | 111 | 124 | 121
Participants | 6 | 4 | 3 | 12

31. Secondary Outcome: Number of Participants Infected With Parasites With the Mutation Pfcrt 76T on Day 0 of the Initial Episode of Malaria
Description: The presence of parasites with the mutation pfCRT 76T was measured with filter paper specimens collected at the time of enrollment and with successful parasite DNA amplification using pyrosequencing.
Time Frame: Day 0 of initial episode of malaria
Population: All participants from whom samples were successfully collected and DNA successfully amplified were included.
Measure: Number; unit: participants
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 159 | 159 | 159 | 158
participants | 1 | 0 | 0 | 0

32. Secondary Outcome: Number of Participants Infected With Parasites With the Mutation Pfcrt 76T at Recrudescent Episodes of Malaria
Description: Participants were enrolled in the study at the time of the initial episode of malaria. If the participant presented with a subsequent episode of malaria at any time during the one year of follow-up, the presence of parasites with the mutation pfCRT 76T was measured with filter paper specimens collected at the time of enrollment and with successful parasite DNA amplification using pyrosequencing.
Time Frame: Recrudescent episodes of malaria within one year of enrollment
Population: The analysis population is limited to participants who presented with subsequent episodes of malaria from whom samples were successfully collected and DNA successfully amplified.
Measure: Number; unit: participants
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 75 | 70 | 74 | 63
participants | 0 | 0 | 1 | 0

33. Secondary Outcome: Number of Participants With New and Recrudescent Malaria Infections After Initial Treatment
Description: Participants were enrolled at the time of initial malaria episode and treated. Subsequent to treatment, subjects were monitored for the occurrence of new and recrudescent malaria infections, which were distinguished by analysis of the infecting parasites using merozoite surface protein-2 polymorphic gene length variation.
Time Frame: 28 days to 1 year
Population: All subjects completing the initial treatment were included in the analysis population.
Measure: Number; unit: participants
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 155 | 148 | 157 | 151
participants
  New infections | 0 | 0 | 1 | 0
  Recrudescent infections | 1 | 0 | 0 | 0

34. Secondary Outcome: Number of Participants With New and Recrudescent Infections After Subsequent New Episodes
Description: Participants were enrolled at the time of initial malaria episode and treated. Subsequent to treatment, participants who subsequently suffered new malaria episodes were monitored for the additional occurrence of new and recrudescent malaria infections, which were distinguished by analysis of the infecting parasites using merozoite surface protein-2 polymorphic gene length variation.
Time Frame: Day 28 to 1 year
Population: The analysis population is limited to participants who had new episodes of malaria during the follow-up period after treatment.
Measure: Number; unit: participants
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 71 | 64 | 67 | 56
participants
  New infections | 0 | 0 | 1 | 1
  Recrudescent infections | 0 | 0 | 2 | 1

35. Secondary Outcome: Time to First Malaria Episode in Participants Who Travelled and Slept Outside the City Versus Those Who Did Not Travel and Sleep Outside the City.
Description: The cumulative hazard of having a malaria attack within one year for those participants who travelled and slept in rural areas (outside the city) versus those who did not was calculated and is presented as a life table to display the number of subjects at risk, the number with first clinical episode and the number censored at each time point. Participants are right-censored at the time of first malaria episode. Participants who did not develop malaria during follow-up or were lost to follow-up were censored at the time of their last visit.
Time Frame: Days 0 - 420
Measure: Number; unit: participants
Groups:
- Participants Who Traveled and Slept Outside the City: At enrollment, participants were asked if they travelled and slept outside the city within the previous 4 weeks. This group indicated yes.
- Participants Who Did Not Travel and Sleep Outside the City: At enrollment, participants were asked if they travelled and slept outside the city within the previous 4 weeks. This group indicated no.
Arm/Group | Participants Who Traveled and Slept Outside the City | Participants Who Did Not Travel and Sleep Outside the City
Number analyzed (Participants) | 432 | 201
participants
  Days 0-27 - Number At Risk | 432 | 201
  Days 0-27 - Number with Malaria | 0 | 0
  Days 0-27 - Number Censored | 63 | 28
  Days 28-55 - Number At Risk | 369 | 173
  Days 28-55 - Number with Malaria | 13 | 4
  Days 28-55 - Number Censored | 26 | 10
  Days 56-83 - Number At Risk | 330 | 159
  Days 56-83 - Number with Malaria | 11 | 9
  Days 56-83 - Number Censored | 21 | 16
  Days 84-111 - Number At Risk | 298 | 134
  Days 84-111 - Number with Malaria | 12 | 12
  Days 84-111 - Number Censored | 16 | 10
  Days 112-139 - Number At Risk | 270 | 112
  Days 112-139 - Number with Malaria | 13 | 4
  Days 112-139 - Number Censored | 17 | 5
  Days 140-167 - Number At Risk | 240 | 103
  Days 140-167 - Number with Malaria | 3 | 2
  Days 140-167 - Number Censored | 22 | 7
  Days 168-195 - Number At Risk | 215 | 94
  Days 168-195 - Number with Malaria | 3 | 1
  Days 168-195 - Number Censored | 16 | 3
  Days 196-223 - Number At Risk | 196 | 90
  Days 196-223 - Number with Malaria | 4 | 4
  Days 196-223 - Number Censored | 16 | 9
  Days 224-251 - Number At Risk | 176 | 77
  Days 224-251 - Number with Malaria | 12 | 1
  Days 224-251 - Number Censored | 4 | 6
  Days 252-279 - Number At Risk | 160 | 70
  Days 252-279 - Number with Malaria | 12 | 1
  Days 252-279 - Number Censored | 8 | 5
  Days 280-307 - Number At Risk | 140 | 64
  Days 280-307 - Number with Malaria | 7 | 4
  Days 280-307 - Number Censored | 4 | 3
  Days 308-335 - Number At Risk | 129 | 57
  Days 308-335 - Number with Malaria | 8 | 5
  Days 308-335 - Number Censored | 8 | 2
  Days 336-363 - Number At Risk | 113 | 50
  Days 336-363 - Number with Malaria | 8 | 3
  Days 336-363 - Number Censored | 2 | 7
  Days 364-391 - Number At Risk | 103 | 40
  Days 364-391 - Number with Malaria | 2 | 0
  Days 364-391 - Number Censored | 100 | 38
  Days 392 - 420 - Number At Risk | 1 | 2
  Days 392 - 420 - Number with Malaria | 0 | 0
  Days 392 - 420 - Number Censored | 1 | 2
Statistical Analysis 1: Comparison: Participants Who Traveled and Slept Outside the City vs Participants Who Did Not Travel and Sleep Outside the City; Test type: Superiority or Other; p = 0.79, Regression, Cox — Not adjusted, 0.05; There are no adjustments; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.68 to 1.34], Standard Error of Mean 0.17 — The reference category is those who did not travel

36. Secondary Outcome: Nearest Neighbor Index as a Measure of Spatial Pattern of the Distribution of Malaria Cases in Ndirande
Description: The Global Positioning System (GPS) was used to establish the coordinates of participants' homes. The distribution of these coordinates was analyzed for evidence of clustering, or occurring closer together than would be expected on the basis of chance. Nearest Neighbor Index is a ratio of the observed mean distance over the expected mean distance. If the index is less than 1, the pattern exhibits clustering. If the index is greater than 1, the trend is toward dispersion.
Time Frame: 1 year
Population: The analysis included all participants for whom the GPS coordinates of the home were established.
Measure: Number; unit: Index
Groups:
- All Groups: Participants Receiving Any Treatment in the Study
Arm/Group | All Groups
Number analyzed (Participants) | 343
Index | 0.328

37. Secondary Outcome: Pharmacokinetics of Chloroquine Represented by Time of Maximal Concentration (Tmax) and Chloroquine Half-life
Description: 1727 non-zero concentration measurements from 479 participants were pooled and used for population pharmacokinetic modeling in Monolix413s. Compartmental population pharmacokinetic modeling was used due to highly sparse data. The model was parameterized in terms of absorption rate constant for chloroquine (Ka), apparent clearance for chloroquine (CL/F, with F as the unknown oral bioavailability), apparent volume of distribution of the central and peripheral compartments for chloroquine (Vd/F), and the inter-compartmental clearance for chloroquine (Q/F). Only these primary population pharmacokinetic parameters could be estimated using the type of data collected. The best-fit population PK model was then used to estimate individual parameter estimates to derive Tmax and half-life.
Time Frame: Day 0 - Day 28
Population: All participants with non-zero concentration measures suitable for pharmacokinetic analysis were included.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 125 | 118 | 120 | 116
Hours
  Time of maximal concentration (Tmax) | 5.6 [5.5 to 5.6] | 5.6 [5.5 to 5.7] | 5.5 [5.4 to 5.5] | 5.6 [5.5 to 5.7]
  Chloroquine half-life | 41.6 [39.4 to 45.7] | 46.2 [43.1 to 48.6] | 41.3 [39.3 to 43.2] | 44.5 [41.0 to 46.8]

38. Secondary Outcome: Pharmacokinetics of Chloroquine Represented by Maximum Concentration (Cmax)
Description: 1727 non-zero concentration measurements from 479 participants were pooled and used for population pharmacokinetic modeling in Monolix413s. Compartmental population pharmacokinetic modeling was used due to highly sparse data. The model was parameterized in terms of absorption rate constant for chloroquine (Ka), apparent clearance for chloroquine (CL/F, with F as the unknown oral bioavailability), apparent volume of distribution of the central and peripheral compartments for chloroquine (Vd/F), and the inter-compartmental clearance for chloroquine (Q/F). Only these primary population pharmacokinetic parameters could be estimated using the type of data collected. The best-fit population PK model was then used to estimate individual parameter estimates to derive Cmax in nanograms per milliliter (ng/mL).
Time Frame: Day 0 - Day 28
Population: All participants with non-zero concentration measures suitable for pharmacokinetic analysis were included.
Measure: Median (95% Confidence Interval); unit: ng/mL chloroquine
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Number analyzed (Participants) | 125 | 118 | 120 | 116
ng/mL chloroquine | 351.0 [295.7 to 388.5] | 345.1 [283.5 to 386.1] | 353.1 [310.6 to 399.1] | 384.2 [309.4 to 394.6]

ADVERSE EVENTS:
Time Frame: Participants were evaluated for adverse events every four weeks through one year after enrollment.
Arm/Group | Chloroquine Plus Artesunate | Chloroquine Plus Atovaquone-Proguanil | CQ Plus Azithromycin | CQ Monotherapy
Serious Adverse Events (participants affected / at risk) | 8/160 | 14/160 | 7/160 | 20/160
Other Adverse Events (participants affected / at risk) | 144/160 | 140/160 | 143/160 | 145/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chloroquine Plus Artesunate (N=160) | Chloroquine Plus Atovaquone-Proguanil (N=160) | CQ Plus Azithromycin (N=160) | CQ Monotherapy (N=160)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral malaria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
HIV infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kwashiorkor (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Febrile convulsion (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Elective surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chloroquine Plus Artesunate (N=160) | Chloroquine Plus Atovaquone-Proguanil (N=160) | CQ Plus Azithromycin (N=160) | CQ Monotherapy (N=160)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 26 (32) | 28 (32) | 32 (36) | 38 (41)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 8 (8) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (11) | 6 (6) | 6 (6) | 5 (6)
Conjunctivitis (Eye disorders) | 27 (29) | 19 (21) | 31 (39) | 31 (38)
Abdominal pain (Gastrointestinal disorders) | 12 (15) | 8 (9) | 16 (20) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 42 (53) | 25 (33) | 26 (33) | 35 (49)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 5 (5) | 5 (5) | 14 (14)
Vomiting (Gastrointestinal disorders) | 4 (4) | 7 (7) | 11 (11) | 7 (8)
Pyrexia (General disorders) | 31 (35) | 22 (22) | 29 (31) | 28 (30)
Body tinea (Infections and infestations) | 14 (14) | 10 (10) | 9 (10) | 6 (6)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3) | 5 (5) | 11 (11)
Conjunctivitis bacterial (Infections and infestations) | 2 (2) | 2 (2) | 7 (7) | 9 (9)
Dysentery (Infections and infestations) | 17 (24) | 8 (8) | 12 (14) | 11 (14)
Gastroenteritis (Infections and infestations) | 46 (53) | 38 (41) | 34 (39) | 40 (44)
Helminthic infection (Infections and infestations) | 8 (8) | 11 (12) | 21 (22) | 10 (11)
Impetigo (Infections and infestations) | 46 (61) | 42 (62) | 31 (37) | 44 (56)
Nasopharyngitis (Infections and infestations) | 128 (358) | 114 (297) | 120 (340) | 119 (335)
Oral herpes (Infections and infestations) | 8 (9) | 5 (5) | 2 (2) | 4 (4)
Otitis media (Infections and infestations) | 12 (12) | 11 (18) | 11 (13) | 15 (20)
Parotitis (Infections and infestations) | 8 (8) | 1 (1) | 4 (4) | 7 (7)
Pneumonia (Infections and infestations) | 36 (50) | 18 (23) | 29 (39) | 40 (50)
Tinea capitis (Infections and infestations) | 23 (27) | 10 (11) | 14 (17) | 14 (15)
Varicella (Infections and infestations) | 17 (17) | 11 (11) | 5 (5) | 16 (16)
Excoriation (Injury, poisoning and procedural complications) | 10 (10) | 6 (6) | 6 (6) | 6 (6)
Thermal burn (Injury, poisoning and procedural complications) | 9 (9) | 7 (7) | 5 (5) | 6 (6)
Alanine aminotransferase increased (Investigations) | 6 (6) | 4 (4) | 10 (10) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (31) | 28 (36) | 28 (32) | 30 (37)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 23 (25) | 32 (34) | 21 (23)
Rash papular (Skin and subcutaneous tissue disorders) | 18 (20) | 24 (26) | 20 (21) | 19 (20)
Rash pruritic (Skin and subcutaneous tissue disorders) | 9 (10) | 4 (4) | 4 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less